CLINICAL TRIAL: NCT05571618
Title: A Multicenter, Real-world Study of the Efficacy and Safety of Antibody-drug Conjugates (ADCs) Rechallenge in Patients with Prior Exposure to ADCs Metastatic Breast Cancer
Brief Title: The Rechallenge of ADCs in MBC Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-23
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Antibody-drug conjugates; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group1
  Interventions: Drug: ADC

INTERVENTIONS:
Drug: ADC — Patients with prior exposure to ADC (either in the adjuvant setting or metastatic disease are allowed).

SUMMARY:
To investigate the efficacy and safety of ADC rechallenge

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old.
* Diagnosed with Metastatic Breast Cancer.
* Patients with prior exposure to ADC (either in the adjuvant setting or metastatic disease are allowed).
* Patients plan to or have received ADCs for the second or more time.
* Complete medical history was available.

Exclusion Criteria:

* Medical history was incomplete

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
ORR | 6 weeks
  Objective Response Rate
CBR | 6 weeks
  Clinical Benefit Rate
DoR | 6 weeks
  Duration of Response
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
OS | 6 weeks
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided